CLINICAL TRIAL: NCT04326686
Title: Examining Factors Influencing Adherence to and Efficacy of a Wholegrains and Nuts Intervention to Reduce Blood Pressure in Prehypertension: a Series of N-of-1 Interventional Studies
Brief Title: Measuring Individual Responses to a Wholegrains and Nuts Intervention to Reduce Blood Pressure in Prehypertension
Acronym: MI-DIET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MI-DIET
Record Dates: First submitted 2020-03-20; First posted 2020-03-30 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Prehypertension
Keywords: N-of-1; Ecological Momentary Assessment; Blood pressure; Whole grains; Nuts
MeSH Terms: conditions — Prehypertension | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: This is a series of N-of-1 studies where data from each participant will be analysed separately. Each study follows an A1-B-A2 design consisting of an initial observation phase, an intervention phase and a follow-up phase, each of 8 weeks duration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N-of-1 study (Other): For 24 weeks, each participant will measure their blood pressure and respond to questionnaires daily, and visit the institute to provide a blood sample every 4 weeks. The study is split into three 8-week phases, the first of which will start when each participant is enrolled. For the first 8-week observation phase (A1) the participant is instructed to continue with their usual diet and exercise habits. For the second 8-week intervention phase (B), the participant will be provided with wholegrains and nuts and recommended to substitute these in place of refined grains and other snacks, respectively. They will also receive dietary advice for following the Dietary Approaches to Stop Hypertension (DASH) diet. For the final 8 week follow-up period (A2), provision of wholegrains and nuts will cease but the participant will continue with measurements at the same frequency as previously.
  Interventions: Other: Dietary intervention: nuts and wholegrains with dietary advice for a blood-pressure lowering diet

INTERVENTIONS:
Other: Dietary intervention: nuts and wholegrains with dietary advice for a blood-pressure lowering diet — 30g mixed unsalted tree nuts (almonds, hazelnuts and almonds) per day; 3 portions of wholegrain foods per day (including wholegrain cereal products, wholegrain bread and wholegrain pasta); guidance for following the Dietary Approaches to Stop Hypertension (DASH) diet

SUMMARY:
The aim of the study is to investigate whether physiological, psychological and environmental factors, at an individual level, modify a) adherence, and b) blood pressure response, to a nuts and wholegrains intervention in participants at risk for developing high blood pressure. For 24 weeks, participants will, on a daily basis, monitor their own blood pressure using a wireless blood pressure monitor and respond to short semi-personalised questionnaires using a wrist-worn device, which also measures activity levels. Participants will receive an intervention of wholegrain foods and nuts to substitute into their diets for 8 weeks, between two 8-week observation periods. The length of the study periods will enable repeated measurements to be taken, in order to assess what factors, on an individual level, are associated with fluctuations in the outcomes. This will provide an insight into the types of factors that can help to explain individual fluctuations in adherence and physiological outcomes, such as blood pressure, that are common in nutrition studies. In the future, this should help in tailoring the way the investigators deliver effective individualised interventions, and enable researchers to be better able to consider and control for factors that can affect adherence and response to dietary interventions.

DETAILED DESCRIPTION:
The study will be conducted as an interventional N-of-1 study with an A1-B-A2 design of 8 weeks per study period. Prior to the study, participants will be screened and if eligible, will complete a number of baseline questionnaires to provide an overview of their typical eating and lifestyle-related behaviours, and general health. A second visit prior to the start of the study will then be arranged, where participants will undergo a semi-structured interview. Responses from the interview, in combination with their baseline questionnaire responses, will be used to identify factors specific to the participant that show some degree of variability. These will form the basis of the semi-personalised questionnaires delivered via the wrist-worn PRO-Diary device for the duration of the study. During the study, participants will visit the institute in a fasted state every 4 weeks (7 visits total), in order to provide a blood sample for assessment of cholesterol levels and for assessment of biomarkers of wholegrains intake. At the first visit, participants will receive the wireless blood pressure monitor and PRO-Diary wrist device programmed with twice-daily questionnaires at times convenient to the participant. After 2 weeks and every 4 weeks thereafter, participants will be sent a link by email to complete a 24-hour dietary recall. After 8 weeks, participants will begin the intervention phase and receive wholegrains equivalent to 3 portions a day and 1 portion of unsalted nuts per day for the following 8 weeks. Participants will be able to choose from a variety of wholegrain products commonly available at supermarkets. They will also receive dietary advice to follow a Dietary Approaches to Stop Hypertension (DASH) diet aimed at lowering blood pressure. All other measures will continue as previously. At week 16, the wholegrains and nuts will be withdrawn and participants will be followed up for a further 8 weeks. At their final visit to the institute, they will complete the same validated questionnaires as at baseline. Results from the study will be analysed using N-of-1 dynamic modelling to analyse trends over time and determine whether any personalised factors significantly affected adherence to intervention or blood pressure response.

ELIGIBILITY:
Inclusion Criteria:

* Mildly elevated blood pressure levels: systolic blood pressure (SBP) >120 <=140mmHg and/or diastolic blood pressure (DBP) >80 <=90mmHg.
* Low habitual intake of wholegrains: <=7 portions/week
* Body Mass Index (BMI) between 18-35
* Possessing a smartphone capable of running the Qardio app in conjunction with the QardioArm wireless blood pressure monitor

Exclusion Criteria:

* SBP <120 or >140mmHg or DBP <80 or >90mmHg. Participants with SBP > 140 or DBP > 90 will be advised to visit their GP to have their blood pressure reassessed in a clinical setting.
* Diagnosed with diabetes
* Clinically diagnosed with hypertension or hypercholesterolemia
* Unstable or untreated thyroid disorder
* Taking blood pressure- or cholesterol-lowering medications (e.g. beta blockers or statins)
* Following a low carbohydrate/gluten free diet
* Coeliac disease/gluten insensitivity
* Any food allergies
* Being on a weight loss diet or having lost >5kg in the last 6 months
* Any history of an eating disorder
* >7 portions/week habitual wholegrains consumption
* Having taken part in a study where wholegrains were provided in the last 3 months
* Not possessing a smartphone to run the Qardio app.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Adherence to wholegrains and nuts consumption | 8-week intervention period
  Number of portions of wholegrains consumed and whether a portion of nuts were consumed, reported daily via the PRO-Diary wrist device.
Change in plasma alkylresorcinol levels reflecting wholegrains intake | Every 4 weeks from start of study up to 24 weeks
  Concentration of alkylresorcinols as a measure of wholegrains intake in nmol/L
Change in blood pressure | From start of study up to 24 weeks
  Blood pressure (both systolic and diastolic) will be taken daily by participants via the QardioArm wireless blood pressure monitor. 3 measurements are taken automatically and averaged.

SECONDARY OUTCOMES:
Correlation between adherence and blood pressure change | 8-week intervention period
  Correlation between adherence and blood pressure change will be examined using N-of-1 dynamic modelling. Daily blood pressure measurements and PRO-Diary questionnaire responses will be provided during the whole study. Questionnaire responses will be given on a Visual Analogue Scale from 0-100.
Total, LDL and HDL cholesterol levels | 4-week blood samples
  Fasted blood samples will be taken to determine whether wholegrains and nuts consumption has an effect on blood cholesterol levels.
Amount of wholegrains and nuts consumed during follow-up reported using PRO-Diary questionnaires | 8-week follow-up phase
  For the final 8 weeks of the study, provision of wholegrains and nuts will cease but participants will continue to be asked about their consumption of these products through daily PRO-Diary questionnaires. This is to determine if habit formation has occurred and led to continuation of consumption of these products
Determination of personal factors which correlate with study outcomes using Ecological Momentary Assessment (EMA) through the PRO-Diary device | 24 weeks
  Participants will respond to semi-personalised questionnaires daily using a Visual Analogue Scale from 0-100 using the PRO-Diary device. The PRO-Diary will also track movement collected during 60-second epochs via accelerometry. The influence of these factors on the primary and secondary outcomes above will be aggregated using N-of-1 dynamic modelling. Due to the semi-personalised nature of the questionnaires, the exact predictors examined in each N-of-1 study will differ. Analysis of each N-of-1 study will be conducted separately.

CONTACTS AND LOCATIONS:
Overall Officials: Baukje de Roos, Principal Investigator — The Rowett Institute, University of Aberdeen
Locations (1):
- The Rowett Institute, University of Aberdeen, Aberdeen, Aberdeen City, United Kingdom

IPD SHARING:
Plan to Share IPD: No